CLINICAL TRIAL: NCT02462161
Title: Study of Nasal Insulin to Fight Forgetfulness - Short-Acting Insulin Aspart
Acronym: SNIFF-Quick
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH); General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00026106; 5P50AG005136-30 (NIH)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Insulin Aspart; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Aspart (Experimental): Fifteen randomly assigned participants with Alzheimer's disease or mild cognitive impairment will receive twice daily intranasal administrations of insulin aspart (20 IU) for 12 weeks.
  Interventions: Drug: Insulin aspart
- Placebo (Placebo Comparator): Fifteen randomly assigned participants with Alzheimer's disease or mild cognitive impairment will receive twice daily intranasal administrations of placebo (saline) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin aspart — Participants will administer 20 IU insulin aspart two times per day with an intranasal delivery device.
  Other Names: NovoLog Fast-Acting Insulin Aspart
  Arms: Insulin Aspart
Drug: Placebo — Participants will administer placebo two times per day with an intranasal delivery device.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This pilot clinical trial will examine the effects of intranasal insulin aspart on cognition, daily function, blood and cerebral spinal fluid markers of Alzheimer's disease, and amyloid deposition in the brain. Participants will be randomly assigned to receive insulin aspart or placebo during a 12-week treatment period.

DETAILED DESCRIPTION:
A growing body of evidence suggests that insulin plays a role in normal memory processes and that insulin abnormalities may contribute to cognitive and brain changes associated with Alzheimer's disease (AD). Interestingly, insulin administered to the nasal cavity is transported within a few minutes into the brain, but does not affect blood sugar or insulin levels.

This trial will consist of a randomized double-blind, placebo-controlled parallel group trial in which 30 participants with AD or mild cognitive impairment (MCI) receive twice daily intranasal administrations of insulin aspart (20 IU) or placebo (saline), two times per day for 12 weeks. All participants will appoint a "support person" to answer a collateral questionnaire and supervise the administration of the study drug. All participants and study partners will undergo the intensive, structured training program in the self-management of intranasal insulin administration. Cognitive testing and blood collection will occur at baseline, after 6 weeks of treatment, and at the end of the 12 week treatment period. Participants will also receive a lumbar puncture to measure AD biomarkers in the subject's cerebral spinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Previous or subsequent diagnosis of Alzheimer's disease or mild cognitive impairment
* Ability to communicate in English

Exclusion Criteria:

* Preexisting diabetes
* Clinically significant elevations in liver function test
* Clinically significant elevations in lipid profile
* Prior lumbar lumbar surgeries or other medical conditions that render lumbar punctures unsafe
* Hemoglobin <8 g/dl
* Significant neurologic disease that might affect cognition, other than Alzheimer's disease, including stroke, Parkinson's disease, multiple sclerosis, or recent severe head injury (within the last year) with loss of consciousness >30 minutes or with permanent neurologic sequelae
* Significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease
* Current use of antipsychotic, anticonvulsant, anxiolytic, anticoagulant or sedative medications
* Current or previous use of glucose-lowering agents or insulin;
* Chronic use (≥ 3 times per week) of nasal sprays of any type for any indication
* Premenopausal status (defined as having had a period within the last year).

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Change in cognition | 6 weeks and 12 weeks
  Alzheimer's Disease Assessment Scale-Cognitive Subscale(ADAS-Cog)/mild cognitive impairment (MCI) scores and memory composite (summed Z scores from delayed story and list recall)

SECONDARY OUTCOMES:
Cerebral spinal fluid (CSF) and blood amyloid-beta, tau protein, and inflammatory markers | Blood - every 6 weeks for 12 weeks; cerebral spinal fluid (CSF) - baseline and week 12
MRI measure of cortical thickness in Alzheimer's disease (AD) -vulnerable regions | Baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT02462161/ICF_000.pdf